CLINICAL TRIAL: NCT05900427
Title: A Double-Blind Randomized Comparison Trial of Postoperative Pain in Patients Undergoing Total Shoulder Arthroplasty Who Receive Interscalene Blocks With or Without Liposomal Bupivacaine (PoPTSAWoW Trial)
Brief Title: Effects on Postoperative Pain of Liposomal Bupivacaine in Interscalene Blocks for Total Shoulder Arthroplasty Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johnny K. Lee (Other)
Collaborators: Endeavor Health (Other)
Responsible Party: Sponsor-Investigator, Johnny K. Lee, M.D., FPA, Principal Investigator, Endeavor Health
Organization: Endeavor Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EH23-069
Record Dates: First submitted 2023-05-22; First posted 2023-06-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Total Shoulder Arthroplasty; Reverse Total Shoulder Arthroplasty
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivacaine Group (Experimental): 10 mL (133 mg) Liposomal bupivacaine and 20 mL (50 mg) 0.25% bupivacaine and 6 mL of saline (183 mg)
  Interventions: Drug: Liposomal bupivacaine
- Plain Bupivacaine Group (Other): 36 mL (180 mg) 0.5% bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Subjects randomized to the Liposomal bupivacaine group will receive 10 mL (133 mg) of Liposomal bupivacaine and 20 mL (50 mg) of 0.25% bupivacaine and 6 mL of saline (183 mg).
  Other Names: Exparel
  Arms: Liposomal Bupivacaine Group
Drug: Bupivacaine — Subjects randomized to the Plain Bupivacaine group will receive 36 mL (180 mg) of 0.5% bupivacaine.
  Other Names: Marcaine
  Arms: Plain Bupivacaine Group

SUMMARY:
The purpose of this trial is to compare the difference in the proportion of patients with tolerable pain scores, VAS pain scores, quality of recovery and opioid use in milligram equivalents (at 24, 48, 72, 96 and 120 hours postoperatively) in patients undergoing shoulder arthroplasty who receive interscalene blocks with or without Liposomal Bupivacaine.

This is a prospective randomized, double-blinded, controlled trial that will enroll 130 subjects undergoing total shoulder arthroplasty or reverse total shoulder arthroplasty. Participants who meet all eligibility criteria will be randomized in a 1:1 ratio to receive either 36 mL of 0.5% bupivacaine (PB group) or 10 mL of liposomal bupivacaine and 20 mL of 0.25 % bupivacaine and 6 mL of saline (LB group).

DETAILED DESCRIPTION:
Patients undergoing shoulder surgery can suffer from significant postoperative pain which can lead to an increase in recovery time, opioid use and potential dependency, and a decrease in quality of recovery. The interscalene brachial plexus block is a common effective regional anesthesia technique used for a variety of procedures involving the shoulder. The number of total shoulder arthroplasty surgeries being performed annually in the United States are increasing every year. Liposomal bupivacaine was FDA approved for use in patients undergoing interscalene block in 2018 to reduce postoperative pain from shoulder surgery. The information from the manufacturer indicates that the liposomal encapsulation may release the drug for up to approximately 72 hours after it has been administered, providing a prolonged analgesic effect. Evidence to the prolonged analgesic effect of liposomal bupivacaine has varied in the current literature. A recent meta-analysis suggested that liposomal bupivacaine may provide a statistically significant, but clinically insignificant decrease in opioid consumption and pain scores over time. The authors noted a possible limitation of their study is that the meta-analysis included a variety of surgical procedures and block techniques, and was not specific to shoulder surgery or interscalene block. The authors noted that this variability in anesthetic regimens between study groups could have affected the observed outcomes.

Recently, the investigators performed a retrospective quality improvement study to investigate the potential benefit of liposomal bupivacaine used for interscalene blocks among 491 patients undergoing shoulder arthroplasty between 2018 and 2021. The investigators compared the difference in the proportion of patients with clinically tolerable pain scores (defined as VAS ≤ 4) in those patients receiving liposomal bupivacaine vs. those receiving another local anesthetic (plain bupivacaine, mepivacaine or ropivacaine) vs. those receiving no block. The results of this study suggested there was significant difference in the proportion of patients with clinically tolerable pain scores when receiving liposomal bupivacaine during all observations and at 3 days postoperatively versus those patient that did not. The patients who received liposomal bupivacaine also had a significant reduction in morphine milligram equivalents (MMEs).

Based on the investigators retrospective results, the investigators performed a power analysis which allowed for the development of this prospective randomized double blinded trial comparing liposomal bupivacaine plus plain bupivacaine vs. plain bupivacaine only in near equipotent doses. The investigators believe that this is a very important and unique trial to perform as it could change the way pain management is delivered in this patient population. Longer acting local anesthetic used for interscalene blocks may increase the number of patients who have tolerable pain and require less or no opioids. This could reduce or inevitably eliminate the unwanted effects of opioids (nausea, vomiting, constipation, urinary retention, opioid induced respiratory depression, dependency and addiction) and result in an improvement in the quality of recovery of patients undergoing total shoulder arthroplasties.

ELIGIBILITY:
Inclusion Criteria:

* Subject ages 18-90 years old
* Male or Female subjects
* Weight ≥ 60 kg.
* Must be able to consent in English

Exclusion Criteria:

* Ages: <18 and >90
* Weight < 60 kg
* Multiple surgeries during one hospital stay
* Emergency surgery
* Allergy or any contraindication to local anesthetics used in trial.
* Pregnancy
* Contraindicated for use of liposomal bupivacaine
* Severe liver/kidney disease
* Defined as a diagnosis of end-stage renal disease (ESRD) defined as being on dialysis
* Subject who received another local anesthetic block prior to the interscalene block.
* Unable to consent in English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The difference in the proportion of patients with clinically significant tolerable pain scores | at Post-operative Day 1
  The investigators will collect the difference in the proportion of patients with clinically significant tolerable pain scores (defined as Visual Analogue Scale (VAS) ≤ 4) post-op Day One in those patients receiving an interscalene block with liposomal bupivacaine with plain bupivacaine vs. plain bupivacaine. Subjects will rate their pain level on a scale of 0-10. Number "0" indicates no pain and number "10" indicates terrible pain.

SECONDARY OUTCOMES:
The difference in the proportion of clinical tolerable pain scores in each group | on Post-operative Day 2, Day 3, Day 4, and Day 5
  The investigators will collect the difference in the proportion of clinical tolerable pain scores (defined as Visual Analogue Scale (VAS) ≤ 4) in each group. Subjects will rate their pain level on a scale of 0-10. Number "0" indicates no pain and number "10" indicates terrible pain.
The difference in Visual Analogue Scale (VAS) pain scores (0 - 10) | Upon Post Anesthesia Care Unit (PACU) admission; Day 0; Post-operative Day 1, Day 2, Day 3, Day 4, and Day 5.
  The investigators will collect the difference in VAS pain scores (0 - 10) in each group. Subjects will rate their pain level on a scale of 0-10. Number "0" indicates no pain and number "10" indicates terrible pain.
The difference in quality of recovery survey-15 responses | on Post-operative Day 1, Day 2, Day 3, Day 4 and Day 5.
  The investigators will collect the difference in quality of recovery survey-15 responses in each group. QoR15 survey has a scale of 0-10. Number "0" indicates none of the time and number "10" indicates all of the time.
Opioid use in morphine milligram equivalents (MME) | on day of surgery; on Post-operative Day 1, Day 2, Day 3, Day 4, and Day 5
  The investigators will collect opioid use in morphine milligram equivalents data from the patients electronic medical record and via an electronic survey sent to patients.
Use of non-opioid analgesics | on day of surgery; on Post-operative Day 1, Day 2, Day 3, Day 4, and Day 5
  The investigators will collect the use of non-opioid analgesics data from the patients electronic medical record and via an electronic survey sent to patients.
Adverse Block Event Survey | on Post-operative Day 1, Day 2, Day 3, Day 4, Day 5 and Day 30
  The investigators will monitor patients for any adverse reaction to the interscalene block by distributing an electronic survey.

CONTACTS AND LOCATIONS:
Overall Officials: Johnny K Lee, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Skokie, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

REFERENCES:
- [Background] Lee HY, Kim SH, So KY, Kim DJ. Effects of interscalene brachial plexus block to intra-operative hemodynamics and postoperative pain for arthroscopic shoulder surgery. Korean J Anesthesiol. 2012 Jan;62(1):30-4. doi: 10.4097/kjae.2012.62.1.30. Epub 2012 Jan 25. PMID 22323951
- [Background] Mirza F, Brown AR. Ultrasound-guided regional anesthesia for procedures of the upper extremity. Anesthesiol Res Pract. 2011;2011:579824. doi: 10.1155/2011/579824. Epub 2011 May 30. PMID 21716734
- [Background] Best MJ, Aziz KT, Wilckens JH, McFarland EG, Srikumaran U. Increasing incidence of primary reverse and anatomic total shoulder arthroplasty in the United States. J Shoulder Elbow Surg. 2021 May;30(5):1159-1166. doi: 10.1016/j.jse.2020.08.010. Epub 2020 Aug 26. PMID 32858194
- [Background] Gorfine SR, Onel E, Patou G, Krivokapic ZV. Bupivacaine extended-release liposome injection for prolonged postsurgical analgesia in patients undergoing hemorrhoidectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2011 Dec;54(12):1552-9. doi: 10.1097/DCR.0b013e318232d4c1. PMID 22067185
- [Background] Hussain N, Brull R, Sheehy B, Essandoh MK, Stahl DL, Weaver TE, Abdallah FW. Perineural Liposomal Bupivacaine Is Not Superior to Nonliposomal Bupivacaine for Peripheral Nerve Block Analgesia. Anesthesiology. 2021 Feb 1;134(2):147-164. doi: 10.1097/ALN.0000000000003651. PMID 33372953
- [Background] Elmer DA, Coleman JR, Renwick CM, Amato PE, Werner BC, Brockmeier SF, Slee AE, Hanson NA. Comparing bupivacaine alone to liposomal bupivacaine plus bupivacaine in interscalene blocks for total shoulder arthroplasty: a randomized, non-inferiority trial. Reg Anesth Pain Med. 2023 Jan;48(1):1-6. doi: 10.1136/rapm-2022-103997. Epub 2022 Oct 19. PMID 36261261
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725